CLINICAL TRIAL: NCT05005403
Title: A Global First-in-Human Study in NSCLC, HNSCC and Solid Tumors With Azirkitug (ABBV-514) as a Single Agent and in Combination With Budigalimab or Bevacizumab
Brief Title: Study to Assess Adverse Events and Pharmacokinetics in Adult Participants With Non-Small Cell Lung Cancer (NSCLC), Head and Neck Squamous Cell Carcinoma (HNSCC) and Other Solid Tumors, Receiving Intravenous (IV) Infusion of Azirkitug (ABBV-514) Alone or in Combination With Budigalimab or Bevacizumab
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M21-410
Record Dates: First submitted 2021-08-12; First posted 2021-08-13 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Micro Satellite Stable Colorectal Cancer; Gastric/Esophageal Cancer; High-Grade Serous Ovarian Cancer; Pancreatic Cancer; Triple Negative Breast Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Head and Neck Squamous Cell Carcinoma; HNSCC; Solid Tumors; Budigalimab; ABBV-181; ABBV-514; Micro Satellite Stable Colorectal Cancer; MSS-CRC, Gastric Cancer; Esophageal Cancer; GEA; GEJ; High-Grade Serous Ovarian Cancer; HGSOC; Pancreatic Cancer, PDAC; Triple Negative Breast Cancer; TNBC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Esophageal Neoplasms; Pancreatic Neoplasms; Triple Negative Breast Neoplasms; Stomach Neoplasms; Anophthalmia with pulmonary hypoplasia | interventions — budigalimab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (14):
- Part 1 Dose Escalation: Azirkitug (ABBV-514) (Experimental): Participants will receive Azirkitug (ABBV-514).
  Interventions: Drug: Azirkitug
- Part 1 Dose Escalation: Azirkitug (ABBV-514) + Budigalimab (Experimental): Participants will receive Azirkitug (ABBV-514) in combination with budigalimab.
  Interventions: Drug: Azirkitug; Drug: Budigalimab
- Part 2 Dose Expansion: Azirkitug (ABBV-514) (Experimental): Participants will receive Azirkitug (ABBV-514) at recommended dose determined in Dose Escalation portion.
  Interventions: Drug: Azirkitug
- Part 2 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab (Experimental): Participants will receive Azirkitug (ABBV-514) at recommended dose determined in Dose Escalation portion in combination with budigalimab.
  Interventions: Drug: Azirkitug; Drug: Budigalimab
- Part 3 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab (Experimental): Participants will receive Azirkitug (ABBV-514) at recommended dose determined in Dose Escalation portion in combination with budigalimab.
  Interventions: Drug: Azirkitug; Drug: Budigalimab
- Part 4 Dose Expansion: Azirkitug (ABBV-514) (Experimental): Participants will receive Azirkitug (ABBV-514) at recommended dose determined in Dose Escalation portion.
  Interventions: Drug: Azirkitug
- Part 4 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab (Experimental): Participants will receive Azirkitug (ABBV-514) at recommended dose determined in Dose Escalation portion in combination with budigalimab.
  Interventions: Drug: Azirkitug; Drug: Budigalimab
- Part 5 Dose Expansion: Azirkitug (ABBV-514) (Experimental): Participants will receive Azirkitug (ABBV-514) at recommended dose determined in Dose Escalation portion.
  Interventions: Drug: Azirkitug
- Part 5 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab (Experimental): Participants will receive Azirkitug (ABBV-514) at recommended dose determined in Dose Escalation portion in combination with budigalimab.
  Interventions: Drug: Azirkitug; Drug: Budigalimab
- Part 6 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab (Experimental): Participants will receive Azirkitug (ABBV-514) at recommended dose determined in Dose Escalation portion in combination with budigalimab.
  Interventions: Drug: Azirkitug; Drug: Budigalimab
- Part 7 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab (Experimental): Participants will receive Azirkitug (ABBV-514) at recommended dose determined in Dose Escalation portion in combination with budigalimab.
  Interventions: Drug: Azirkitug; Drug: Budigalimab
- Part 8 Dose Escalation: Azirkitug (ABBV-514) + Bevacizumab (Experimental): Participants will receive Azirkitug (ABBV-514) in combination with bevacizumab.
  Interventions: Drug: Azirkitug; Drug: Bevacizumab
- Part 8 Dose Expansion: Azirkitug (ABBV-514) + Bevacizumab (Experimental): Participants will receive Azirkitug (ABBV-514) at recommended dose determined in Dose Escalation portion in combination with bevacizumab.
  Interventions: Drug: Azirkitug; Drug: Bevacizumab
- Part 9 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab (Experimental): Participants will receive Azirkitug (ABBV-514) at recommended dose determined in Dose Escalation portion in combination with budigalimab.
  Interventions: Drug: Azirkitug; Drug: Budigalimab

INTERVENTIONS:
Drug: Azirkitug — Intravenous (IV) Infusion
  Other Names: ABBV-514
Drug: Budigalimab — Intravenous (IV) Infusion
  Other Names: ABBV-181
  Arms: Part 1 Dose Escalation: Azirkitug (ABBV-514) + Budigalimab; Part 2 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab; Part 3 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab; Part 4 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab; Part 5 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab; Part 6 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab; Part 7 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab; Part 9 Dose Expansion: Azirkitug (ABBV-514) + Budigalimab
Drug: Bevacizumab — Intravenous (IV) Infusion
  Arms: Part 8 Dose Escalation: Azirkitug (ABBV-514) + Bevacizumab; Part 8 Dose Expansion: Azirkitug (ABBV-514) + Bevacizumab

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. Non-Small Cell Lung Cancer (NSCLC) is a solid tumor, a disease in which cancer cells form in the tissues of the lung. Head and Neck Squamous Cell Carcinoma (HNSCC) is a solid tumor, a disease in which cancer cells form in the tissues of the head and neck. The purpose of this study is to assess adverse events and pharmacokinetics of Azirkitug (ABBV-514) as a monotherapy and in combination with Budigalimab or Bevacizumab,.

Bevacizumab is an approved product, while Budigalimab and Azirkitug (ABBV-514) are investigational drugs being developed for the treatment of NSCLC, HNSCC, and other solid tumors. Study doctors put the participants in groups called treatment arms. The maximum-tolerated dose (MTD)/maximum administered dose (MAD) of Azirkitug (ABBV-514) will be explored. Each treatment arm receives a different dose of Azirkitug (ABBV-514) in monotherapy and in combination with Budigalimab or Bevacizumab. Approximately 512 adult participants will be enrolled in the study across approximately 80 sites worldwide.

Participants will receive Azirkitug (ABBV-514) as a monotherapy or in combination with Budigalimab or Bevacizumab as an Intravenous (IV) Infusion for an estimated treatment period of up to 2 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Pre Treatment biopsy or archive tissue within 6 months without intervening treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of <=1
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST)
* Laboratory values meeting criteria outlined in the protocol
* NSCLC - Advanced or metastatic progressed on standard of care (SOC) including chemotherapy and prior anti-PD-(L)1 antibody (separately or in combination). Actionable gene alterations are eligible if failed targeted therapeutic options.
* HSNCC - Advanced/metastatic progressed on platinum and PD-1/PD-LI in recurrent or metastatic setting.
* Micro Satellite Stable Colorectal Cancer (MSS-CRC) - Progressed on Oxaliplatin, Irinotecan, a fluoropyrimidine, anti-EGFR, VEGF or VEGFR therapies, TAS-102, Regorafenib and not MSI-h or MMR-deficient
* Gastric and Gastroesophageal Junction adenocarcinoma (GEA) - Advanced/metastatic progressed on at least 1 prior cytotoxic chemotherapeutic regimen and if applicable immune checkpoint inhibitor and/or HER2 therapy
* High-Grade Serous Ovarian Cancer (HGSOC) - Progressed serous epithelial ovarian, fallopian tube or primary peritoneal cancer post SOC and not eligible for surgical resection. Platinum resistant cannot have >5 lines of prior therapy.
* Pancreatic Adenocarcinoma (PDAC) - Advanced/metastatic progressed after SOC. Includes adenosquamous carcinoma and post-Whipple.
* Triple Negative Breast Cancer (TNBC) - Progressed after >1 systemic therapy that must have included taxane and treatment naïve to immunotherapy targeting T-cell co-stimulation

Exclusion Criteria:

* Pancreatic Ductal Adenocarcinoma (PDAC) - Excludes neuroendocrine or acinar pancreatic carcinoma and participants with coagulopathy or at risk of or history of Deep vein thrombosis (DVT)/PE
* No major surgery within 28 days prior to dosing
* No active autoimmune/immunodeficiency disease with limited exceptions
* Combination treatment excludes participants treated with anti-programmed cell death protein 1(PD-1)/Programmed cell death ligand 1 (PD-L1) who had immune mediated toxicity G3 or greater, interstitial lung disease, or hypersensitivity Combination treatment may also require no significant cardiac deficiencies and/or events
* Pregnancy
* Excluded medications include anticancer therapy within 5 half-live or 28 days (whichever is shorter), agent targeting Chemokine Receptor (CCR)8, live vaccines, immunosuppressive medication with limited exceptions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE) | Up to 2 Years
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Serum Concentration (Cmax) of ABBV-514 | Up to 2 Years
  Maximum Observed Serum Concentration (Cmax) of of ABBV-514.
Time to Maximum Observed Serum Concentration (Tmax) of ABBV-514 | Up to 2 Years
  Time to maximum Observed Serum Concentration (Tmax) of of ABBV-514.
Terminal Elimination Half-Life (t1/2) of ABBV-514 | Up to 2 Years
  Terminal elimination half-life (t1/2) of ABBV-514.
Area Under the Serum Concentration Versus Time Curve (AUC) of ABBV-514 | Up to 2 Years
  Area under the serum concentration versus time curve (AUC) of ABBV-514.
Antidrug Antibody (ADA) | Up to 2 Years
  Incidence and concentration of anti-drug antibodies.
Neutralizing Antidrug Antibody (nADA) | Up to 2 Years
  Incidence and concentration of neutralizing anti-drug antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (35):
- United States (14):
  - City of Hope National Medical Center /ID# 276272, Duarte, California
  - University of Illinois Hospital and Health Sciences System /ID# 251750, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc /ID# 232593, Fort Wayne, Indiana
  - Community Health Network, Inc. /ID# 243011, Indianapolis, Indiana
  - Norton Cancer Institute /ID# 248903, Louisville, Kentucky
  - START Midwest /ID# 248685, Grand Rapids, Michigan
  - Nebraska Cancer Specialists - Omaha - Wright Street /ID# 247399, Omaha, Nebraska
  - Carolina BioOncology Institute /ID# 232597, Huntersville, North Carolina
  - NEXT Oncology Austin /ID# 243005, Austin, Texas
  - The University of Texas MD Anderson Cancer Center /ID# 270059, Houston, Texas
  - NEXT Oncology /ID# 243007, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics (START) /ID# 276268, San Antonio, Texas
  - Start Mountain Region /ID# 276270, West Valley City, Utah
  - Virginia Cancer Specialists - Fairfax /ID# 232592, Fairfax, Virginia
- Israel (4):
  - The Chaim Sheba Medical Center /ID# 238332, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 238333, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 252287, Jerusalem
  - Rabin Medical Center /ID# 250497, Petah Tikva
- Japan (7):
  - Aichi Cancer Center Hospital /ID# 250405, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 238840, Kashiwa-shi, Chiba
  - Kobe University Hospital /ID# 250409, Kobe, Hyōgo
  - Kansai Medical University Hospital /ID# 276805, Hirakata-shi, Osaka
  - Shizuoka Cancer Center /ID# 250408, Sunto-gun, Shizuoka
  - National Cancer Center Hospital /ID# 238372, Chuo-ku, Tokyo
  - Wakayama Medical University Hospital /ID# 276806, Wakayama, Wakayama
- South Korea (5):
  - National Cancer Center /ID# 252290, Goyang-si, Gyeonggido
  - CHA Bundang Medical Center /ID# 252291, Seongnam, Gyeonggido
  - Yonsei University Health System Severance Hospital /ID# 252288, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 252289, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 252867, Seoul, Seoul Teugbyeolsi
- Taiwan (5):
  - National Taiwan University Hospital /ID# 251894, Taipei City, Taipei
  - Taipei Medical University Shuang Ho Hospital /ID# 252449, New Taipei City
  - National Cheng Kung University Hospital /ID# 252262, Tainan
  - Taipei Medical University Hospital /ID# 252450, Taipei
  - Tri-Service General Hospital /ID# 252263, Taipei

IPD SHARING:
Plan to Share IPD: No